CLINICAL TRIAL: NCT03001024
Title: WayToServe Español: A Culturally-Appropriate Online Responsible Beverage Service Training for Spanish-Speaking Servers
Brief Title: WayToServe Español: Online Responsible Beverage Service Training for Spanish-Speaking Servers
Acronym: WTS-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: University of Texas, El Paso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R44MD010405-03 (NIH); 0311 (Other: Klein Buendel, Inc.)
Record Dates: First submitted 2016-11-21; First posted 2016-12-22 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Alcoholic Intoxication
MeSH Terms: conditions — Alcoholic Intoxication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation of WayToServe Español (Experimental): The experimental design to be employed in the trial evaluation of WayToServe Español (WTS-E) in this direct-to-Phase II project is a two-arm randomized field trial design (WTS-E vs. Usual and Customary [UC] training) with three assessment points (pretest - immediate post-test - 9 month follow-up).This constitutes a 2 (level of RBS training intervention) x 3 (level of time assessment) mixed factorial design. Spanish dominant onsite and off-site licensed alcohol premises will be the unit of analysis, stratified by type of premise (onsite vs. off-site sales) and state (New Mexico vs. Texas).
  Interventions: Behavioral: Implementation of WayToServe Español
- Usual and Customary RBS Training (Active Comparator): The Investigators have carefully considered the over-time assessment factor in this design, and have chosen two follow-up assessments over a 9 month-period because a) our prior WayToServe® trials have shown that an immediate post-training assessment will document intervention effects when training effects are at optimum levels immediately after the training; b) the sustained effect of WTS-E needs to be demonstrated to show long-term not just short-term impact (9 months being between our previous 6-month and 1-year follow-ups). Finally, c) all follow-ups can be completed within the approximately 2-year period of a Phase II project. The immediate post-training assessment will occur for both arms of the design, one month after premises in the intervention arm are given access to WTS-E.
  Interventions: Behavioral: Usual and Customary RBS Training

INTERVENTIONS:
Behavioral: Implementation of WayToServe Español — Following baseline assessment and randomization to experimental condition, premises assigned to the intervention condition will be contacted and recruited to the trial. Managers will provide a list of all servers. All servers will be registered by project staff on the WTS-E website and provided a unique identification code, which will track their use of the training and associate it with the premise. Servers will complete a profile on the program during their first login. Servers will be asked to complete the training within four weeks from initial registration; email and text reminders will be sent to those who do not login within one week of initial registration.
  Arms: Implementation of WayToServe Español
Behavioral: Usual and Customary RBS Training — The premises randomized to the UC training condition will be, in effect, blind to the investigation. Server training is mandatory for all servers in New Mexico. Server training is voluntary in Texas but heavily incentivized by TABC's Safe Harbor clause. Under this clause, liquor licensees are held harmless for any service infractions if all servers are trained and certified by an approved RBS trainer; instead, the server is cited for the infraction.
  Arms: Usual and Customary RBS Training

SUMMARY:
Responsible Beverage Service Training (RBS) has been shown to be effective and recent research by this research team has shown that online RBS training (WayToServe®) was more effective, particularly over time, than usual and customary (UC) RBS training by live trainers. However, one growing segment of alcohol servers and sellers has been neglected in RBS training efforts: Hispanic primarily Spanish-speaking servers in predominantly Spanish-speaking premises. This project will develop and test the first online RBS training for predominantly Spanish-speaking servers, WayToServe Español, which is culturally and linguistically appropriate and will fill a gap in evidence-based alcohol prevention interventions for this underserved population.

DETAILED DESCRIPTION:
Among the measures against drunk driving available to policy makers and prevention practitioners, Responsible Beverage Service (RBS) training has shown promise. In these programs, alcohol servers are educated in a number of techniques, including correct identification checking, recognizing signs of intoxication in patrons, and managing patrons via drink counting techniques to safely keep them under Driving While Intoxicated blood alcohol limits. Recent reviews of RBS programs have found evidence for effectiveness. However, the diffusion of RBS training and practices has been limited: 18 U.S. states require some form of RBS training, another 18 incentivize training in some way, and the other 14 states have no RBS regulations at all. As a result, while RBS training may be widely available, it is not widely adopted. An overlooked limitation of all RBS training in the U.S., and a limit to its dissemination, is that it is only offered in English and from a mainstream U.S. culture point of view. Proposed here is the development and testing of a Spanish-language version of an evidence-based online RBS training program (WayToServe®) that will be culturally tailored to Hispanic cultural values, experiences, and circumstances: WayToServe Español. The systematic development of WayToServe Español will meet the training needs of an underserved and growing population segment of alcohol servers and sellers - Hispanics who are predominant speakers of Spanish and who often work in premises with many predominantly Spanish-speaking patrons. The proposed Direct-to-Phase II research will be accomplished in two phases. The first phase will entail the iterative and systematic development of WayToServe Español via Spanish-language focus groups and usability testing. The second phase will involve the evaluation of WayToServe Español in Spanish-dominant premises in New Mexico and West Texas via a randomized efficacy trial that randomly assigns premises to either receive WayToServe Español training or Usual and Customary (UC) RBS training. A variety of alcohol service refusal rates will be the primary outcome variable, measured using a pseudo-intoxicated Pseudo-Patron (PP) buyer assessment protocol. Premises will be assessed at baseline, post-training, and 9-month follow up intervals. Should WayToServe Español prove effective, commercialization plans include efforts similar to those for WayToServe® (English), now available in four states (New Mexico, Texas, California, Washington, and under review for approval in Oregon) and having trained nearly 29,000 alcohol servers and sellers. Overall, the project will bolster efforts to diffuse an effective RBS training to underserved Spanish-speaking alcohol servers and sellers, benefitting both them directly and the communities in which they live. WayToServe Español will be the first culturally- and linguistically-appropriate evidence-based RBS training available online in the U.S. for this underserved population.

ELIGIBILITY:
Inclusion Criteria:

* Speak Spanish Primarily or bilingual in Spanish and English
* Serve alcohol in a Spanish-dominant premise in New Mexico or West Texas
* Age 18 or older

Exclusion Criteria:

* Have a family member who is participating in the project
* Speak English primarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Alcohol Service Refusal | 9 Months
  The Investigators will employ data forms completed by both PP buyer and observer to record server reactions during the PP buyer visit. These forms are filled out immediately after the visit and are checked by research staff for completeness and concordance before data entry. The PP buyer form contains fields that record if an alcohol sale was made. The alcohol service refusal rate is the ratio of the number of times the sale is refused to the number of purchase attempts.

SECONDARY OUTCOMES:
Effect Moderator - Physical Layout/Decor of the Establishment | 9 Months
  Descriptive data about the physical layout/decor of the premises
Effect Moderator - Approximate Number of Servers On Duty | 9 Months
  Data about the approximate number of servers on duty
Effect Moderator - Approximate number of patrons | 9 Months
  Data about the approximate number of patrons in establishment
Effect Moderator - Gender of Server Who Interacts with PP buyer | 9 Months
  Data about the gender of server who interacts with PP buyer
Effect Moderator - Approximate Age of Server Who Interacts with PP Buyer | 9 Months
  Data about the approximate age of server who interacts with PP buyer
Effect Moderator - Server and PP buyer Interaction - Duration | 9 Months
  Data about the duration of the alcohol service request
Effect Moderator - Server and PP Buyer Interaction - Server Comments | 9 Months
  Descriptive data about comments from server
Effect Moderator - Server and PP Buyer Interaction - Server Interference | 9 Months
  Descriptive data about the attempts by server to intervene and not serve
Effect Moderator - Onsite or Off-site Premise | 9 Months
  Data regarding if premise is onsite vs. off-site
Effect Moderator - New Mexico or Texas | 9 Months
  Data regarding if premise is located in New Mexico or Texas

CONTACTS AND LOCATIONS:
Overall Officials: Gill Woodall, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Klein Buendel, Inc., Golden, Colorado
  - University of Texas, El Paso, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No